CLINICAL TRIAL: NCT06890676
Title: Extending Infection Control Dental Care to Nursing Home Residents Using Telehealth-Mediated Supervision: a Novel Solution to Nursing Home Acquired Pneumonia Morbidity and Mortality.
Brief Title: Extending Dental Care to Nursing Home Residents to Reduce Mouth Infections and Incidence of Pneumonia and Improve Diabetic Glucose Control
Acronym: NHOralHealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Missouri Department of Health and Senior Services (Other)
Responsible Party: Principal Investigator, Guy Deyton, Project Specialist, Missouri Department of Health and Senior Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-0501; T1246090 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis; Gingivitis; Periodontal Disease; Periodontal Infections; Oral Infections; Periapical Infections; Pneumonia; Diabetes
Keywords: Nursing Home; Long-Term Care Facility; Dental Care; Dental Infections; Oral Infections; Periodontal Infections; Periodontal Diseases; Dental Caries; Pneumonia; Diabetes; Oral Hygiene; Caries Arrest; Frailty; Telehealth
MeSH Terms: conditions — Periodontitis; Gingivitis; Periodontal Diseases; Pneumonia; Diabetes Mellitus; Dental Caries; Frailty | interventions — Periodontal Debridement; Tooth Exfoliation; Root Planing; Fluoride Treatment; Toothbrushing; Referral and Consultation; Drainage; Anti-Infective Agents; Tooth Extraction

STUDY DESIGN:
Masking Description: The Primary investigator and Outcomes Assessor are blinded to the identities of the patients and facilities. The data will be pooled and considered in affregate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infection Control Arm (Experimental): * Dental Hygienists and EFDA Teams travel to nursing homes and gather medical and dental data for residents participating in the study while collaborating with distant dentists using telehealth.
  * Clinical data is sent to the supervising dentist, who reviews medical history, assigns an ASA class and Frailty class, and prescribes an infection control treatment plan.
  * Emergent infections outside the scope of hygienists / EFDAs result in a transport order for care to an outside facility.
  * Hygienist/EFDA teams treat residents in their facility for gum infections, stabilize decay with fluoride and temporary fillings, and clean dentures.
  * The hygienist/EFDA team teaches LTCF staff oral hygiene assistance techniques to help residents with daily care and minimize reinfection.
  * The hygienist and EFDA team will continue to see LTCF residents at regular intervals to provide maintenance care, collect data, and monitor progress.
  * Treatment Outcome Data collected.
  Interventions: Other: Comprehensive Oral Evaluation; Other: Intraoral Complete Radiographic Series; Other: • Teledentistry-synchronous and asynchronous; Procedure: Periodontal Therapy; Procedure: Periodontal Maintenance Procedure; Procedure: Application of Caries Arresting Medicament; Other: Oral Hygiene Assistance; Procedure: Referral for Treatment of Acute Oral Infection

INTERVENTIONS:
Other: Comprehensive Oral Evaluation — A thorough check-up of teeth, gums, and surrounding tissues, including medical and dental history, to assess overall oral health and identify any infections.
  Other Names: Oral Hygiene Assistance Arm; Data Collection Using Telehealth-Mediated Supervision
Other: Intraoral Complete Radiographic Series — A series of x-rays of the whole mouth intended to display the, teeth, roots, periapical areas, bone, and areas without teeth.
Other: • Teledentistry-synchronous and asynchronous — The delivery or coordination of care for a patient using synchronous; real-time or aysnchronous communication between care providers or between care providers and a patient.
Procedure: Periodontal Therapy — A therapeutic procedure designed to remove plaque and calculus (hardened plaque) causing gum infections that can lead to tooth loss and other medical complications.
  Other Names: Periodontal Debridement; Scaling and Root Planing; Scaling in the Presence of Gingival Inflammation
Procedure: Periodontal Maintenance Procedure — A periodic evaluation and therapeutic support procedure for patients with a history of gum infections.
Procedure: Application of Caries Arresting Medicament — Topical application of decay arresting or inhibiting medicament.
  Other Names: Fluoride Treatment; Silver Diamine Fluoride Treatment
Other: Oral Hygiene Assistance — Dental procedures aimed at educating patients on, and assisting patients with ,proper oral hygiene practices removing food debris, germ-laden plaque, and soft tartar using cloth wipes, toothbrush, floss, and using oral hygiene aids.
  Other Names: Oral Hygiene Instruction; Toothbrushing; Denture Cleaning
Procedure: Referral for Treatment of Acute Oral Infection — Diagnosis and treatment of oral infection outside the scope of a dental hygienist or Expanded Function Dental Assistant.
  Other Names: Incision and Drainage; Antibiotic Therapy; Tooth Extraction

SUMMARY:
The goal of this study is to learn if dental infection control treatment delivered to older adult nursing home residents at their place of residence will result in :

* improved dental health
* reduced risk of pneumonia
* better glucose control for diabetic patients compared to the pre-project dental and general health evaluations of residents and the pre-project facility incidence of pneumonia. Dental infection control treatment includes treating gum infections, stopping or slowing decay with fluoride, and assisting residents with effective tooth brushing and denture cleaning daily. Previous studies indicate dental infections can be inhaled and cause pneumonia or make diabetes worse. A shortage of dentists has limited care for nursing home residents. This project will allow dental hygienists and specially trained dental assistants to treat nursing home residents using telehealth methods (computers, cameras, internet, and telephone) to talk and work with dentists in different locations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the periodontal health of nursing home residents who receive dental infection control treatment at their residential nursing care facility provided by dental hygienists and dental assistants compared to the pre-project health evaluations of the same patients using diagnostic criteria endorsed jointly by the American Academy of Periodontists and the European Federation of Periodontists.

SECONDARY OBJECTIVES II. To evaluate the incidence of pneumonia in the group of nursing home residents who received dental infection control treatment 1 year after treatment compared to the facility incidence of pneumonia for the same period preceding the start of the dental care project.

III. To evaluate the level of glucose control of diabetic nursing home residents for 1 year after they received dental infection control compared to glucose control of the same diabetic nursing home residents before receiving the treatment using serum HbA1c sampling.

IV. To evaluate the effectiveness of an oral hygiene assistance mentoring program for nursing home staff to improve the oral hygiene of the nursing residents using a simple resident oral hygiene evaluation instrument administered by visiting dental hygienists.

V. To evaluate the effectiveness of an oral hygiene assistance mentoring program for nursing home staff to increase their knowledge about oral hygiene and the relationship between oral infections and systemic disease using pre-course and post-course comprehension tests.

VI. To evaluate the effectiveness of decay stabilization treatment using topically applied fluoride and SMART fillings delivered to nursing home residents by hygienists and dental assistants compared to residents who do not receive such care using physical inspection and dental radiographs.

VII. To evaluate the effectiveness of using near-infrared imaging function of a continuous intraoral scan to evaluate decay stabilization treatment using topically applied fluoride and SMART fillings delivered to nursing home residents by hygienists and dental assistants compared to traditional dental radiographs and physical inspection using Likert surveys of attending dentists.

VIII. To evaluate the effectiveness of a novel frailty assessment instrument, the Modified Frail Questionnaire, as a screening instrument to discriminate nursing home residents who can be safely treated by hygienists and assistants in their residential facility using a Lickert Scale evaluation survey of attending dentists and by reporting adverse incidents encountered during the project.

IX. To evaluate the perceived value of this dental care program by residents and/or family members using Lickert Scale evaluations X. To evaluate the perceived value of the dental care program by nursing home staff using Likert Scale evaluations.

XI. To evaluate the perceived sustainability of the dental care program by dental contractors using Likert Scale evaluations.

Outline: Dental contractors were recruited by published RFA and attended an in-person workshop outlining study requirements, nursing home facility recruitment, participant informed consent process, and data submission requirements. Contractors met with nursing home facilities, educated them about the project, and enlisted staff assistance to recruit study participants from the census of residents of participating nursing homes. Residents were interviewed, educated, screened for inclusion and exclusion, and serially admitted to the study with signed consent for participation, dental infection control treatment, and access to their medical records.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 60 years of age residing in a nursing home or communal care setting;
* Review of Medical history results in an assigned American Society of Anesthesiologists Physical Status Evaluation of Class II or III;
* Frailty Assessment of Low or Moderate using the Modified FRAIL Questionnaire;
* Consent is required for study participation, disease control oral healthcare, and access to medical records.

Exclusion Criteria:

* Age < 60;
* American Society of Anesthesiologists Physical Status Evaluation of Class IV or V;
* High frailty evaluation using the Modified FRAIL Questionnaire;
* Resident deemed behaviorally or physically difficult to treat by initial clinical assessment.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Periodontal Health | One year from the delivery of the infection control interventional care
  I. To evaluate the periodontal health of nursing home residents who receive dental infection control treatment compared to their pre-treatment peroidontal assessment using periodontal probe and inflammation diagnostic criteria endorsed by the American Academy of Periodontists and the European Federation of Periodontists.

SECONDARY OUTCOMES:
Pneumonia Incidence | One year from the delivery of the infection control interventional care
  To evaluate the incidence of pneumonia in the group of nursing home residents who received dental infection control treatment compared to the facility incidence of pneumonia preceding the start of the dental care project.
Diabetic Glucose Control | One year from the delivery of the infection control interventional care
  To evaluate the level of glucose control of diabetic nursing home residents for 1 year after they received dental infection control treatment compared to glucose control of the same diabetic nursing home residents before receiving the treatment using serum HbA1c sampling
Oral Hygiene Assistance Instruction | One year from the delivery of the infection control interventional care
  To evaluate the effectiveness of an oral hygiene assistance mentoring program for nursing home staff to improve the oral hygiene of the nursing residents using 'Hygienist Assessment of Resident Oral Hygiene' administered by visiting dental hygienists. This instrument rates oral hygiene on a scale of 1 (poor) to 5 (good). The individual scores will be reported as aggregate scores monthly using mean and standard deviation comparing resident oral hygiene.
Decay Stabilization Treatment | One year from the delivery of the infection control interventional care#
  VI. To evaluate the effectiveness of decay stabilization treatment using topically applied fluoride and SMART fillings delivered to nursing home residents by hygienists and dental assistants compared to residents pre-treatment evaluation of untreated decay using physical inspection, dental radiographs, and infra-red decay detection. The individual treatment evaluations will be recorded in REDCap 6 and 12 month after treatment and summarized in aggregate in a table entitle: 'Outcomes of Decay Stabilization Treatment in Nursing Home Residents'. The outcome fields of the table are: # untreated/unstable Decayed teeth at Initial Examination; # untreated/unstable Decayed Teeth at 6 Month Evaluation; # untreated/unstable Decayed Teeth at Final Evaluation; % Change in Untreated/Unstable Decayed Teeth.
Frailty Assessment | One year from the delivery of the infection control interventional care
  To evaluate the effectiveness of the Modified Frail Questionnaire as a screening instrument using a Likert Scale evaluation survey of attending dentists and by reporting adverse incidents encountered during the project. The Modified Frail Questionnaire evaluates five criteria: fatigue, resistance, ambulation, illnesses, and weight loss, yielding a 0 or 1 score for each category. Total category scores of 0 or 1 = low frailty; 2-3 = moderate frailty; 4-5 = high frailty. Attending dentists assess the effectiveness of the Frailty Questionnaire using a Likert Evaluation entitled: 'Supervising Dentist Assessment of the Modified Frail Questionnaire as a Risk Assessment Instrument' with 1 indicating a very low level of satisfaction and 10 indicating a very high level of satisfaction. Adverse incidents are reported using a protocol-prescribed form and will be reported in the discussion portion of the project report.
Patient's / Families' Perceived Value of Dental Program | One year from the delivery of the infection control interventional care.
  To evaluate the perceived value of this dental care program by residents and/or family members using Likert Scale evaluation entitled: 'Patient / Guardian assessment of Oral Healthcare Program in Residential Care Facilities'. The instrument uses a 1 t0 10 scale with 1 indicating a very low level of satisfaction and 10 indicating a very high level of satisfaction.
Nursing Home Staff Perceived Value of Dental Program | One year from the delivery of the infection control interventional care
  To evaluate the perceived value of the dental care program by nursing home staff using Likert Scale evaluation entitled 'LTCF Staff Assessment of Oral Healthcare Program in Residential Care Facilities'. The instrument uses a 1 to 10 scale with 1 with 1 indicating a very low level of satisfaction and 10 indicating a very high level of satisfaction.
Dental Contractor Perceived Sustainability of Dental Program | One year from the delivery of the infection control interventional care.
  To evaluate the perceived sustainability of the dental care program by dental contractors using Likert Scale evaluation entitled: 'Contractor Assessment of Feasibility & Sustainability of Project'. This instrument uses a 1 to 10 scale with 1 indicating a low level of sustainability and significant barriers to sustainability and 10 being a high level of sustainability with few barriers to sustain the project.

CONTACTS AND LOCATIONS:
Locations (1):
- Office of Dental Health, Department of Health and Senior Services, Jefferson City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed in aggregate to ensure the confidentiality of each study participant and the facilities involved in the study

REFERENCES:
- See also: MedlinePlus: What is Pneumonia? — https://medlineplus.gov/pneumonia.html